CLINICAL TRIAL: NCT03694093
Title: A Prospective Study Assessing the Effect of Patient Characteristics on Treatment Response in Hyperhidrosis
Brief Title: Assessing the Effect of Patient Characteristics on Treatment Response in Primary Hyperhidrosis
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Dee Anna Glaser, MD, Interim Chair, Department of Dermatology, St. Louis University
Other Study IDs: 29446
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Hyperhidrosis: Subjects with Primary Hyperhidrosis will be followed in this study. Because this study is observational, there will be no intervention.

SUMMARY:
This study will describe the treatment of hyperhidrosis (excessive sweating) in clinical practice and explore the effect of patient characteristics on treatment response. This study will follow 200 people with hyperhidrosis over 18 months. Anyone with primary hyperhidrosis (excessive sweating not due to another medical condition) over the age of 12 may participate. Study participants will have multiple office visits during which they will asked to rate the severity of their sweat production in multiple areas (i.e. underarms, hands, feet), answer a questionnaire regarding their disease and treatment, and undergo a non-invasive measurement of sweat production called gravimetry. Gravimetry is performed by placing absorbent material in an area, such as the underarms, for a set amount of time and then measuring the amount of sweat collected. In between clinic visits, study participants will be contacted electronically to answer several questions regarding their disease and treatment.

DETAILED DESCRIPTION:
Subject Recruitment

Recruitment will take place at SLUCare Dermatology Des Peres Clinic. Patients with non-study related appointments with Dr. Glaser regarding the management of primary hyperhidrosis will be approached by a research member. Patients will be given ample time to review study design and have questions and concerns addressed. After inclusion and exclusion criteria, study purpose and design, signed consent (parent or guardian will sign if subject is a minor), assent (for minors only, not signed) and HIPAA release are attained, the patients will be enrolled in the study.

The investigators will be recruiting two types of patients for this study. (1) New patients being seen for evaluation for primary hyperhidrosis. These subjects will be presenting to the hyperhidrosis clinic for the first time. If enrolled, these subjects will have all data prospectively collected. (2) Established patients being seen for ongoing management of primary hyperhidrosis who have documented baseline gravimetric measurements (defined as measurements taken while the patient was undergoing no active therapies for primary hyperhidrosis). These subjects will be presenting to the hyperhidrosis clinic for continued care. If enrolled, these subjects will have some data collected retrospectively with the remainder collected prospectively (see below for details).

Withdrawal or Discontinuation

Subjects may withdraw from the study at any time. If a subject desires withdraw from the study, the subject will be give a reason for study withdraw which will be included in publication. If a subject misses a scheduled visit the subject will be contacted via phone to ask if the subject is withdrawing from the study or reschedule a visit.

Because the subjects are only undergoing gravimetry, a non invasive way of measuring sweat production, it is highly unlikely that there would be any reason to discontinue a subjects participation due to safety. However, if at any point the supervising provider feels that a patient is at risk of harm the subject may be withdrawn from the study. In this case, a reason would be recorded for publication purposes.

Screen Failures

For those that fail screening, all information collected prior to that time will be shredded and disposed of in confidentiality trash bins. Only a reason for failing to pass screening will be recorded for publication purposes.

Subject Visits

Subjects will be screened, sign consent (parent or guardian will sign if subject is a minor), review assent (only applicable to minors) HIPAA release, and enrolled at an initial visit. Patients will have a monthly electronic or telephone survey to fill out. Patients will be seen every 3 months in clinic until the patient has achieved treatment response and/or no treatment changes are required. 6 months after this visit, the patient will be seen in clinic again***. If the subject has a sustained treatment response and/or has no treatment change, the subject will exit the study. If these conditions are not met, then the subject will resume 3 month visits.

It is important to note that these visit will overlap with non-study related visits that occur as a part of management of the patient's disease. Disease management decisions, such as which therapy to prescribe, will occur independently of this study and will not be affected by study participation. All visits will occur within 18 months after the study begins. No further study encounters will occur after this time period regardless of treatment changes or response.

*** Subjects may choose to forgo this 6 months visit and complete it electronically or by telephone.

New Patient

Subject Visit 1, 1 hour:

The subject will first verify his or her name and contact information. After the subject agrees to study participation they will sign a consent (permission) and a release of health information. Consent will be signed by parent or guardian if the subject is a minor. If the subject is a minor assent will also be reviewed with the subject. Inclusion and exclusion criteria will be reviewed.

Through an interview with a research team member and chart review, the following data will be collected:

* Basic demographics
* Current treatments
* Hyperhidrosis Disease Severity Scale score (a scale that rates how the subject feels sweating affects daily activities) for all sites:
* Scalp
* Face
* Underarms
* Inframammary
* Chest
* Back
* Hands
* Feet
* Groin
* Buttocks
* Questionnaire regarding the subject's disease state (see attachment).

Patients will then undergo gravimetric measurements of all sites affected by hyperhidrosis as detailed in the attachment. Areas affected by HH will be defined by areas with an HDSS 3 or greater. For details on the gravimetry protocol, see attachment.

Subject Visits, follow-up, 30 minutes:

The following data will be collected through subject interview:

* Current treatment
* HDSS for all sites.
* Questionnaire regarding the subject's disease state (see attachment).
* Presence or absence of side effects

Patients will then undergo gravimetric measurements for sites with previous measurements. For detailed protocol see attachment.

Established Patient

Subject Visit 1, 1 hour:

The subject will first verify his or her name and contact information. After the subject agrees to study participation they will sign a consent (permission) and a release of health information. Consent will be signed by parent or guardian if the subject is a minor. If the subject is a minor assent will also be reviewed with the subject. Inclusion and exclusion criteria will be reviewed.

Through chart review, the following data will be collected:

* Baseline (defined as data collected while the patient was not undergoing any treatment) HDSS score and gravimetric measurements for all sites
* Number of treatment changes since initiating care
* Basic demographics

Through an interview with the patient, the following information will be collected:

* Current treatment
* HDSS score for all sites
* Questionnaire regarding the subject's disease state (see attachment).
* Presence or absence side effects

Patients will then undergo gravimetric measurements for sites with previous gravimetric measurements.

Subject Visit, follow-up 30 minutes:

This will be the same as new patient follow up visits.

Subject Electronic/Telephone Survey: Monthly, 15 minutes

The following data will be collected through a phone or electronic interview between a research team member and the subject:

- Questionnaire regarding the subject's disease state (see attachment).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race who has received the diagnosis of primary Hyperhidrosis at any site
2. Patients receiving continued treatment of primary Hyperhidrosis with baseline gravimetrics (established patients only) performed at SLUCare Dermatology Des Peres clinic. Baseline gravimetrics are defined as measurements taken during times of no active disease interventions.

Exclusion Criteria:

1. Received the following therapies at the site being evaluated prior to baseline gravimetrics:

   1. Botulinum toxin injections 6 months prior to baseline gravimetric data collection.
   2. Applied Aluminum chloride on day of baseline gravimetric data
   3. Ongoing iontophoresis therapy at time of baseline gravimetric data
   4. Oral systemic anticholinergics 4 weeks prior to baseline gravimetric data
   5. Received surgical intervention, suction and curettage, microwave thermolysis, or ultrasound therapy prior to baseline gravimetrics.
2. Patient has received diagnosis of secondary hyperhidrosis (i.e hyperhidrosis due to an underlying medical condition such as hyperthyroidism)
3. Younger than 12 years of age.
4. Does not desire study participation or is unable to consent.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or Females ≥ 12 with Primary Hyperhidrosis.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Weeks till treatment response | 18 months
  We will measure the weeks required to reach treatment response defined as HDSS of 1 or 2.

SECONDARY OUTCOMES:
Number of treatment changes | 18 months
  We will quantify the number of failed treatment prior to treatment response.
Number of treatments at the time of treatment response. | 18 months
  We will quantify the number of treatments a subject is currently using at the time of treatment response.
Percent reduction in gravimetric sweat measurements | 18 months
  We will quantify the percent reduction in gravimetric sweat measurements from initial visit compared to after treatment response is achieved.
Disease impact | 18 months
  We will track the disease impact through questionnaire responses throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dee A Glaser, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hornberger J, Grimes K, Naumann M, Glaser DA, Lowe NJ, Naver H, Ahn S, Stolman LP; Multi-Specialty Working Group on the Recognition, Diagnosis, and Treatment of Primary Focal Hyperhidrosis. Recognition, diagnosis, and treatment of primary focal hyperhidrosis. J Am Acad Dermatol. 2004 Aug;51(2):274-86. doi: 10.1016/j.jaad.2003.12.029. No abstract available. PMID 15280848
- [Background] Glaser DA, Ballard AM, Hunt NL, Pieretti LJ, Pariser DM. Prevalence of Multifocal Primary Hyperhidrosis and Symptom Severity Over Time: Results of a Targeted Survey. Dermatol Surg. 2016 Dec;42(12):1347-1353. doi: 10.1097/DSS.0000000000000949. PMID 27879523
- [Background] Doolittle J, Walker P, Mills T, Thurston J. Hyperhidrosis: an update on prevalence and severity in the United States. Arch Dermatol Res. 2016 Dec;308(10):743-749. doi: 10.1007/s00403-016-1697-9. Epub 2016 Oct 15. PMID 27744497
- [Background] Basra MK, Fenech R, Gatt RM, Salek MS, Finlay AY. The Dermatology Life Quality Index 1994-2007: a comprehensive review of validation data and clinical results. Br J Dermatol. 2008 Nov;159(5):997-1035. doi: 10.1111/j.1365-2133.2008.08832.x. Epub 2008 Sep 15. PMID 18795920
- [Background] Iwase S, Ikeda T, Kitazawa H, Hakusui S, Sugenoya J, Mano T. Altered response in cutaneous sympathetic outflow to mental and thermal stimuli in primary palmoplantar hyperhidrosis. J Auton Nerv Syst. 1997 Jun 6;64(2-3):65-73. doi: 10.1016/s0165-1838(97)00014-3. PMID 9203126
- [Background] Bovell DL, Clunes MT, Elder HY, Milsom J, Jenkinson DM. Ultrastructure of the hyperhidrotic eccrine sweat gland. Br J Dermatol. 2001 Aug;145(2):298-301. doi: 10.1046/j.1365-2133.2001.04351.x. PMID 11531796
- [Background] Kowalski JW, Eadie N, Dagget S, Lai P-Y. Validity and reliability of the hyperhidrosis disease severity scale (HDSS). J Am Acad Dermatol 2004;50(3):P51.
- [Background] Hoorens I, Ongenae K. Primary focal hyperhidrosis: current treatment options and a step-by-step approach. J Eur Acad Dermatol Venereol. 2012 Jan;26(1):1-8. doi: 10.1111/j.1468-3083.2011.04173.x. Epub 2011 Jul 13. PMID 21749468
- [Background] Benson RA, Palin R, Holt PJ, Loftus IM. Diagnosis and management of hyperhidrosis. BMJ. 2013 Nov 25;347:f6800. doi: 10.1136/bmj.f6800. No abstract available. PMID 24277380
- [Background] Solish N, Bertucci V, Dansereau A, Hong HC, Lynde C, Lupin M, Smith KC, Storwick G; Canadian Hyperhidrosis Advisory Committee. A comprehensive approach to the recognition, diagnosis, and severity-based treatment of focal hyperhidrosis: recommendations of the Canadian Hyperhidrosis Advisory Committee. Dermatol Surg. 2007 Aug;33(8):908-23. doi: 10.1111/j.1524-4725.2007.33192.x. PMID 17661933
- [Background] Wolosker N, Teivelis MP, Krutman M, de Paula RP, de Campos JR, Kauffman P, Puech-Leao P. Long-term results of oxybutynin treatment for palmar hyperhidrosis. Clin Auton Res. 2014 Dec;24(6):297-303. doi: 10.1007/s10286-014-0264-8. Epub 2014 Nov 27. PMID 25427685
- [Background] Wolosker N, Krutman M, Teivelis MP, Paula RP, Kauffman P, Campos JR, Puech-Leao P. Analysis of oxybutynin treatment for hyperhidrosis in patients aged over 40 years. Einstein (Sao Paulo). 2014 Jan-Mar;12(1):42-7. doi: 10.1590/s1679-45082014ao2841. PMID 24728245
- [Background] Wolosker N, Krutman M, Campdell TP, Kauffman P, Campos JR, Puech-Leao P. Oxybutynin treatment for hyperhidrosis: a comparative analysis between genders. Einstein (Sao Paulo). 2012 Oct-Dec;10(4):405-8. doi: 10.1590/s1679-45082012000400002. English, Portuguese. PMID 23386077